CLINICAL TRIAL: NCT04757025
Title: Optimization of Intraoperative Ventilation Guided by Electrical Impedance Tomography in Combination With Oxygen Saturation by Pulse Oximetry (SpO2) Versus SpO2 Alone in Obese Patients Undergoing Robotic Assisted Radical Prostatectomy: Prospective Randomized Trial
Brief Title: Intraoperative Electrical Impedance Tomography in Obese Patients Undergoing Robotic Assisted Radical Prostatectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Ester Forastiere, MD, Head of Department of Anaestesiology and Critical Care, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RS1452/20(2443)
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical Impedance Tomography (Experimental): patient monitored by Electrical Impedance Tomography
  Interventions: Device: Electrical Impedance Tomography
- Peripheral arterial Saturation (Active Comparator): patient monitored by Peripheral arterial Saturation alone
  Interventions: Device: Peripheral arterial Saturation

INTERVENTIONS:
Device: Electrical Impedance Tomography — In 27 patients ventilation will be guided with an Electrical Impedance Tomography system
  Arms: Electrical Impedance Tomography
Device: Peripheral arterial Saturation — The ventilation of 27 patients will be guided by Peripheral arterial Saturation alone
  Arms: Peripheral arterial Saturation

SUMMARY:
The primary objective of our study will be verify a possible improvement in arterial oxygenation in the obese patient undergoing robotic-assisted radical prostatectomy if the ventilation will be guided by electrical impedance tomography rather than peripheral saturation alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laparoscopic radical prostatectomy
* BMI ≥ 30 kg/m2

Exclusion Criteria:

* surgery duration < 2 hours
* history of lung diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
The arterial oxygen pressure / fraction of inspired oxygen (pO2 /FiO2) ratio | 16 months
  The primary outcome will be the ratio of arterial oxygen pressure and the fraction of inspired oxygen (pO2 / FiO2 ratio) at the end of the intervention, detected by blood gas analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Regina Elena Cancer Institute, Rome, RM, Italy